CLINICAL TRIAL: NCT03943342
Title: A Multicenter Study of Ibrutinib Resistance Development and Intervention With Venetoclax (Phase II)
Brief Title: Ibrutinib and Venetoclax in Treating Patients With Chronic Lymphocytic Leukemia After Ibrutinib Resistance
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not feasible
Sponsor: Kerry Rogers (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Kerry Rogers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18311; NCI-2019-02511 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Chronic Lymphocytic Leukemia; Loss of Chromosome 17p
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, ibrutinib) (Experimental): OBSERVATION COHORT: Patients who are taking ibrutinib enter observation cohort and undergo screening every 3 months for development for genetic mutations. If mutations develop, patients undergo increased screening for development of clinical disease progression. Patients who develop clinical disease progression with or without mutations enter the Intervention cohort.
  INTERVENTION COHORT: Patients receive venetoclax PO daily and ibrutinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve MRD negative CR after 12 or 24 cycles continue receiving ibrutinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta

SUMMARY:
This phase II trial studies how well the combination of ibrutinib and venetoclax works in treating patients with chronic lymphocytic leukemia whose cancer has stopped responding to ibrutinib alone. Both ibrutinib and venetoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving ibrutinib and venetoclax together after development of ibrutinib resistance may work better than discontinuing ibrutinib and switching to other chemotherapy drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Overall response rate to combination ibrutinib and venetoclax after 12 cycles (intervention cohort).

II. Rate of mutation negative status after 12 cycles of combination venetoclax and ibrutinib (intervention cohort ).

SECONDARY OBJECTIVES:

I. Incidence of BTK C481S mutations during ibrutinib treatment (observation cohort).

II. Progression-free survival after development of a BTK C481S mutation (observation cohort).

III. Progression-free and overall survival after adding venetoclax to ibrutinib (intervention cohort).

IV. Type and incidence of adverse events during combination ibrutinib and venetoclax treatment in this patient population (intervention cohort).

EXPLORATORY OBJECTIVES:

I. Determine patient and disease characteristics associated with clinical disease progression in a univariable and multivariable analysis (observation cohort).

II. Determine the changes in the allelic frequency of ibrutinib resistance mutations after their development (observation cohort) and after venetoclax is added (intervention cohort).

III. Determine novel resistance mechanisms to ibrutinib and ibrutinib/venetoclax combination therapy by whole exome and ribonucleic acid (RNA) sequencing at baseline and clinical relapse.

IV. Perform BH3 profiling and correlate with response to combination venetoclax and ibrutinib therapy.

OUTLINE: This is a dose-escalation study of venetoclax.

OBSERVATION COHORT: Patients who are taking ibrutinib enter Observation cohort and undergo screening every 3 months for development for genetic mutations. If mutations develop, patients undergo increased screening for development of clinical disease progression. Patients who develop clinical disease progression with or without mutations enter the Intervention cohort.

INTERVENTION COHORT: Patients receive venetoclax orally (PO) daily and ibrutinib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve minimal residual disease (MRD) negative complete remission (CR) after 12 or 24 cycles continue receiving ibrutinib PO QD on days 1-28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic leukemia (CLL) meeting criteria established by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL).
* Currently taking ibrutinib and first took ibrutinib > 12 months ago.
* At high risk for the development of ibrutinib resistance. Patients are considered at high risk for ibrutinib resistance if they have had >= 2 prior therapies for CLL prior to ibrutinib and have either del(17p)(13.1) and/or a complex CLL karyotype.
* Able to continue taking ibrutinib.
* Willing to enter the intervention cohort if clinical disease progression as defined by IWCLL 2018 criteria develops.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Absolute neutrophil count (ANC) >= 1000/mm^3 independent of growth factor support.
* Platelets >= 100,000/mm^3 or >= 50,000/mm^3 if bone marrow involvement independent of transfusion support in either situation.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN).
* Total bilirubin =< 1.5 x ULN unless bilirubin rise is due to Gilbert?s syndrome or of non-hepatic origin.
* Creatinine clearance (CLcr) >30 ml/min.
* Able to take an absorb pill form oral medications.
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.
* CRITERIA FOR ENTERING THE INTERVENTION COHORT: Clinical disease progression as defined by IWCLL 2018 criteria AND presence of an ibrutinib resistance mutation as defined.
* CRITERIA FOR ENTERING THE INTERVENTION COHORT: No evidence of a non-CLL/small lymphocytic lymphoma (SLL) lymphoma (Richter?s syndrome).
* CRITERIA FOR ENTERING THE INTERVENTION COHORT: No contraindication to taking venetoclax.
* CRITERIA FOR ENTERING THE INTERVENTION COHORT: Able to continue taking ibrutinib.

Exclusion Criteria:

* Inability to continue taking ibrutinib for any reason.
* Presence of a known ibrutinib resistance mutation as defined.
* Clinical disease progression while taking ibrutinib as defined by IWCLL 2018 criteria.
* Major surgery or a wound that has not fully healed within 4 weeks of randomization.
* Known central nervous system lymphoma.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon).
* Requires chronic treatment with strong CYP3A inhibitors.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator?s opinion, could compromise the subject?s safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* History of lymphoma (Richter?s syndrome) unless in complete remission > 2 years without relapse.
* History of active malignancies other than CLL within the past 3 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma or the cervix or breast
  * Basal cell or localized squamous cell carcinoma of the skin
  * Previous malignancy treated with curative therapy and not expected to relapse.
* Inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease, etc.).
* Prior allogeneic stem cell transplant with Day 0 < 12 months prior and/or with chronic graft versus host disease (GVHD) requiring current use of immunosuppression. Patients with prior allogeneic stem cell transplant with Day 0 > 12 months prior who do not require immunosuppression for GVHD will be eligible.
* Patients in the observation cohort who develop clinical disease progression and do NOT have a known ibrutinib resistance mutation will be taken off study and may not enter the intervention cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) (intervention cohort) | After 12 cycles of combination therapy, assessed up to 3 years
  Defined as the percentage of patients who have achieved any response better than stable disease after 12 cycles of combination ibrutinib and venetoclax treatment. All eligible patients who take one study dose of venetoclax will be considered evaluable and included in the denominator when calculating the ORR. ORR will be estimated with a 95% exact binomial confidence interval at the response assessment after 12 cycles of combination ibrutinib and venetoclax therapy, and 24 if applicable.
Rate of mutation negative status (intervention cohort) | After 12 cycles of combination therapy, assessed up to 3 years
  Rate of mutation negative status will be estimated with a 95% exact binomial confidence interval at the response assessment after 12 cycles of combination ibrutinib and venetoclax therapy, and 24 if applicable.

SECONDARY OUTCOMES:
Incidence of BTK C481S mutations (observation cohort) | Up to 3 years
  Person-time incidence of developing a BTK C481S mutation will be calculated by dividing the number of new mutations observed while on ibrutinib therapy by the total number of months patients are receiving ibrutinib and were at risk.
Progression-free survival (PFS) after development of a BTK C481S mutation (observation cohort) | Up to 3 years
  Will be calculated in the observation cohort from the date a BTK C481S mutation was first reported until the date of clinical disease progression by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria or death from any cause, whichever occurs first.
PFS after adding venetoclax to ibrutinib (intervention cohort) | Up to 3 years
  PFS will be calculated in the intervention cohort from the start date of combination therapy (C1D1) until the date of progressive disease or death from any cause. Will be described using the method of Kaplan-Meier.
Overall survival (OS) after adding venetoclax to ibrutinib (intervention cohort) | Up to 3 years
  OS will be calculated in the intervention cohort from the start date of combination therapy (C1D1) until the date of progressive disease or death from any cause. Will be described using the method of Kaplan-Meier.
Incidence of adverse events (intervention cohort) | Up to 3 years
  Graded per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 with the exception of hematologic adverse events. Adverse events will be summarized by type, severity and perceived attribution. Hematologic adverse events will be graded according to CLL-specific criteria described in the IWCLL 2018 guidelines. The maximum grade for each type of toxicity will be recorded for each patient and frequency tables will be reviewed to determine the toxicity patterns. In addition, will also summarize the number of patients who discontinue combination therapy due to adverse events.

OTHER OUTCOMES:
Patient and disease characteristics associated with clinical disease progression (observation cohort) | Up to 3 years
  Univariable and multivariable analysis will be performed to determine what patient and disease characteristics are associated with development of ibrutinib resistance mutations. All standard CLL risk characteristics, prior treatments, and standard patient demographic information will be included.
Changes in allelic frequency of ibrutinib resistance mutations after their development (observation cohort) | Up to 3 years
  Univariable and multivariable analysis will be performed to determine what patient and disease characteristics are associated with development of ibrutinib resistance mutations. All standard CLL risk characteristics, prior treatments, and standard patient demographic information will be included.
Changes in allelic frequency of ibrutinib resistance mutations after addition of venetoclax (intervention cohort) | Up to 3 years
  Univariable and multivariable analysis will be performed to determine what patient and disease characteristics are associated with development of ibrutinib resistance mutations. All standard CLL risk characteristics, prior treatments, and standard patient demographic information will be included.
Novel resistance mechanisms to ibrutinib and ibrutinib/venetoclax combination therapy by whole exome and ribonucleic acid (RNA) sequencing (Seq) | At baseline and at clinical relapse, assessed up to 3 years
  For RNA-Seq data analysis, will first use FASTQC for the read quality recalibration, and then conduct removing, trimming, and filtering based on base quality scores and nucleotide distributions. Coverage BED (bedtools package) will be used for counting reads per feature per sample. Filtering of noise level counts across comparison groups will be used to reduce false positives. After filtering, differential expression will be tested using R package limma with voom normalization.
BH3 profiling | Up to 3 years
  Correlate with response to combination venetoclax and ibrutinib therapy. Descriptive statistics such as mean, standard deviation, median, range, etc., for continuous variables and proportions for discrete variables will be used to summarize correlative endpoints in each of the defined strata. Graphical summaries will also be used extensively to visualize the data and describe relationships between variables (e.g. boxplots of BH3 profiling by response status).

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A Rogers, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu